CLINICAL TRIAL: NCT02451124
Title: Office Based Screening Test for Barrett's Esophagus
Brief Title: Non-endoscopic Brushing of the Esophagus Using a Non-endoscopic Inflatable Balloon of the Esophagus in Screening for Barrett Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CASE6214; NCI-2015-00246 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE6214 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH); U54CA163060 (NIH); P50CA150964 (NIH)
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Barrett Esophagus
Keywords: Barrett; Cancer; Screening
MeSH Terms: conditions — Barrett Esophagus; Neoplasms | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening: non-endoscopic inflatable balloon for the esophagus (Experimental): Patients undergo non-endoscopic brushing of the esophagus using a non-endoscopic inflatable balloon for the esophagus over 30-60 minutes followed by a standard esophagogastroduodenoscopy. Questionnaire administration will provide self-reported data on patient experiences. laboratory biomarker analysis of biopsy will confirm diagnosis.
  Interventions: Device: non-endoscopic inflatable balloon for the esophagus; Other: Questionnaire Administration; Other: Laboratory Biomarker Analysis; Procedure: esophagogastroduodenoscopy

INTERVENTIONS:
Device: non-endoscopic inflatable balloon for the esophagus — Undergo non-endoscopic brushing of the esophagus using a non-endoscopic inflatable balloon for the esophagus
  Other Names: Balloon
Other: Questionnaire Administration — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: esophagogastroduodenoscopy — Standard of care, patients digestive tract scoped post balloon brushing
  Other Names: EGD

SUMMARY:
This pilot clinical trial studies non-endoscopic brushing of the esophagus using a non-endoscopic inflatable balloon for the esophagus in screening for Barrett esophagus, a condition where the lining of the esophagus has changed or been replaced with abnormal cells that may lead to cancer. The non-endoscopic inflatable balloon for the esophagus is a capsule balloon that brushes against the walls of the esophagus to collect esophageal samples. Non-endoscopic brushing of the esophagus using a non-endoscopic inflatable balloon for the esophagus may help doctors find Barrett esophagus sooner, when it may be easier to treat.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine acceptability of non-endoscopic balloon brushing of esophagus.

II. To demonstrate successful performance of the methylation of vimentin (mVIM) assay in balloon brushings from subjects with and without Barrett's Esophagus (BE).

III. To examine molecular and histological factors that might lead to false negative and false positive mVIM assays in BE screening.

IV. To assay additional methylated deoxyribonucleic acid (DNA) biomarkers that might improve the sensitivity and specificity of mVIM in balloon brushings.

OUTLINE:

Patients undergo non-endoscopic brushing of the esophagus using a non-endoscopic inflatable balloon for the esophagus over 30-60 minutes followed by a standard esophagogastroduodenoscopy (EGD).

After completion of study, patients with serious adverse events are followed up until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause.

ELIGIBILITY:
Inclusion Criteria:

* Patients are undergoing clinically indicated esophagogastroduodenoscopy (EGD)
* Patients can provide informed consent
* Patients have no known coagulopathy and no known history of esophageal varices

Exclusion Criteria:

* Patients are not undergoing clinically indicated EGD
* Patients have known coagulopathies or history of esophageal varices
* Patients do not have the ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08-11 (Actual); Study Completion 2017-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Chak, Principal Investigator — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Screening: Non-endoscopic Inflatable Balloon for the Esophagus
Started | 156
Completed | 155
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Screening: Non-endoscopic Inflatable Balloon for the Esophagus
Number analyzed (Participants) | 156
Age, Customized [Count of Participants; unit: Participants]
  20-29 | 2
  30-39 | 4
  40-49 | 10
  50-59 | 36
  60-69 | 45
  70-79 | 39
  80-89 | 11
  90-99 | 1
  Unknown | 8
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 48
  Male | 107
  Unknown | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 133
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 126
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 156

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Each Category of Tolerance Assessed by the Tolerance Survey
Description: Mean tolerance score as assessed by 'tolerance survey' with scores ranging from 0 to 50 with higher scores indicating worse tolerance of interventional balloon device. Subscales include anxiety, pain, choking, gagging, and overall tolerance, with each domain scores ranging from 0 to 10, with higher scores indicating worse tolerance of interventional balloon device.
Time Frame: At completion of study procedure (up to 60 minutes)
Population: Participants who were successfully able to swallow the device
Measure: Number; unit: number of participants
Groups:
- Low Discomfort: scores of 1-2 (low discomfort)
- Intermediate Discomfort: Scores of 3-8 (intermediate discomfort)
- High Discomfort: Scores of 9-10 (high discomfort)
Arm/Group | Low Discomfort | Intermediate Discomfort | High Discomfort
Number analyzed (Participants) | 128 | 128 | 128
number of participants
  Anxiety | 96 | 31 | 1
  Pain | 121 | 7 | 0
  Choking | 105 | 22 | 1
  Gagging | 66 | 58 | 4
  Overall tolerance | 92 | 36 | 0

2. Primary Outcome: Sensitivity of the mVIM Assay in Balloon Brushings From Participants With BE
Description: Sensitivity of the mVIM assay in balloon brushings from participants with BE as measured by true positives determined by biomarker (mVIM and mCCNA1) analyses of corresponding esophageal balloon derived samples compared to initial diagnosis. The presence of at least 1% of methylated VIM in DNA extracted from the esophageal sampling balloon will be considered a positive assay.
Time Frame: Up to 1 year
Population: Evaluable Cases. Cases are participants with diagnosed BE. Some cases not evaluable because of failure to swallow device, failure to obtain adequate DNA from balloon tips, or other exclusionary reasons.
Measure: Number; unit: % sensitivity
Groups:
- Screening: Non-endoscopic Inflatable Balloon for the Esophagus: Patients undergo non-endoscopic brushing of the esophagus using a non-endoscopic inflatable balloon for the esophagus over 3-15 minutes followed by a standard EGD. Questionnaire administration will provide self-reported data on patient experiences. laboratory biomarker analysis of biopsy will confirm diagnosis.
  Questionnaire Administration: Ancillary studies
  Laboratory Biomarker Analysis: Correlative studies
  EGD: Standard of care, patients' digestive tract examined with EGD post balloon brushing
Arm/Group | Screening: Non-endoscopic Inflatable Balloon for the Esophagus
Number analyzed (Participants) | 50
% sensitivity | 88

3. Primary Outcome: Specificity of the mVIM Assay in Balloon Brushings From Control Participants With no BE Diagnosis
Description: Specificity of the mVIM assay in balloon brushings from control subjects with BE as measured by true negatives determined by biomarker (mVIM and mCCNA1) analyses of corresponding esophageal balloon derived samples compared to initial control status. The presence of at least 1% of methylated VIM in DNA extracted from the esophageal sampling balloon will be considered a positive assay.
Time Frame: Up to 1 year
Population: Evaluable Controls. Controls were evaluable participants with with no diagnosed disease. Some controls not evaluable because of failure to swallow device, failure to obtain adequate DNA from balloon tips, or other exclusionary reasons.
Measure: Number; unit: % specificity
Arm/Group | Screening: Non-endoscopic Inflatable Balloon for the Esophagus
Number analyzed (Participants) | 36
% specificity | 92

4. Primary Outcome: Average Methylation of Methylated Beta-1,3-glucuronyltransferase 2 Assays
Description: Average methylation of methylated beta-1,3-glucuronyltransferase 2 assays
Time Frame: Up to 7 months
Population: Data not collected
Arm/Group | Screening: Non-endoscopic Inflatable Balloon for the Esophagus
Number analyzed (Participants) | 0

5. Primary Outcome: Performance of the mVIM Assay in Balloon Brushings From Subjects Without BE
Description: Performance of the mVIM assay in balloon brushings from subjects without BE
Time Frame: Up to 7 months
Population: Data not collected
Arm/Group | Screening: Non-endoscopic Inflatable Balloon for the Esophagus
Number analyzed (Participants) | 0

6. Primary Outcome: Average Methylation of Zinc Finger Protein 793 Assay
Description: Average methylation of zinc finger protein 793 assay
Time Frame: Up to 7 months
Population: Data not collected
Arm/Group | Screening: Non-endoscopic Inflatable Balloon for the Esophagus
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: at procedure (average of 24 hours)
Arm/Group | Screening: Non-endoscopic Inflatable Balloon for the Esophagus
All-Cause Mortality (participants affected / at risk) | 0/156
Serious Adverse Events (participants affected / at risk) | 0/156
Other Adverse Events (participants affected / at risk) | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT02451124/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT02451124/Prot_SAP_001.pdf